CLINICAL TRIAL: NCT00055770
Title: A Phase I and Phase II Study of OSI-774 in Combination With Docetaxel in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Erlotinib Plus Docetaxel in Treating Patients With Locally Advanced, Metastatic, or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01432; NCI-2012-01432 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-0213; NCI-5393; CDR0000271197; OSU-02H0084; OSU 0213 (Other: Ohio State University Medical Center); 5393 (Other: CTEP); U01CA076576 (NIH)
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Salivary Gland Squamous Cell Carcinoma; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Docetaxel

ARMS (1):
- Arm I (Experimental): PHASE I: Patients receive oral erlotinib once daily on days 1-28 and docetaxel IV over 1 hour on days 8, 15, and 22. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 6 patients receives erlotinib at the MTD.
  PHASE II: Patients receive erlotinib at the MTD and docetaxel as in phase I.
  Interventions: Drug: erlotinib hydrochloride; Drug: docetaxel; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I/II trial to study the effectiveness of combining erlotinib with docetaxel in treating patients who have locally advanced, recurrent, or metastatic head and neck cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with docetaxel may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and dose-limiting toxicity of erlotinib when administered in combination with docetaxel in patients with locally advanced, metastatic, or recurrent squamous cell carcinoma of the head and neck.

II. Determine the response rate, duration of response, time to progression, and survival of patients treated with this regimen.

III. Determine the pharmacokinetics of this regimen in these patients. IV. Correlate the presence of PTEN, RB, P-Akt, p15, p16, cyclin D1, p27, and p53 genes in tumor tissue with response in patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of erlotinib followed by a phase II study.

PHASE I: Patients receive oral erlotinib once daily on days 1-28 and docetaxel IV over 1 hour on days 8, 15, and 22. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional cohort of 6 patients receives erlotinib at the MTD.

PHASE II: Patients receive erlotinib at the MTD and docetaxel as in phase I.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck meeting 1 of the following staging criteria:

  * Recurrent
  * Metastatic
  * Locally advanced and determined to be incurable by surgery or radiotherapy
* Measurable disease
* No known brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No severe pulmonary insufficiency, including chronic obstructive pulmonary disease, requiring oxygen (O2 saturation less than 90%) and/or increase in PaCO2 blood gas level greater than 50 mm Hg
* No history of abnormality of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Able to take oral medication
* No requirement for IV alimentation
* No active peptic ulcer disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant traumatic injury within the past 21 days
* No prior allergic reactions to compounds of similar chemical or biological composition to study drugs
* No grade 2 or greater persistent peripheral neuropathy
* No other concurrent uncontrolled illness that would preclude study participation
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior immunotherapy for head and neck cancer
* No more than 1 prior chemotherapy regimen in the adjuvant or neoadjuvant setting
* No more than 1 prior chemotherapy regimen for metastatic disease
* No prior docetaxel (phase II only)
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior hormonal therapy for head and neck cancer
* Prior external beam radiotherapy allowed
* At least 4 weeks since prior radiotherapy and recovered
* More than 21 days since prior major surgery
* No prior surgery affecting gastrointestinal absorption
* No prior epidermal growth factor receptor-targeting therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapies or agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of erlotinib and docetaxel, based on incidence of DLT graded according to NCI CTC version 2.0 (Phase I) | Up to 28 days
Proportion of patients with an objective response (Phase II) | Up to 6 years

SECONDARY OUTCOMES:
Response rate as measured by RECIST criteria (Phase II) | Up to 6 years
Time to tumor progression (Phase II) | Up to 6 years
Median survival (Phase II) | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Kraut, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States